CLINICAL TRIAL: NCT05769673
Title: Soft and Hard Tissue Changes Around Implants Using Customized CAD/CAM Healing Abutments
Brief Title: Soft and Hard Tissue Changes Around Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Acela A. Martinez Luna, Clinical Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-000291
Record Dates: First submitted 2023-01-25; First posted 2023-03-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized Healing Abutments (Experimental): Placement of a customized CAD/CAM healing abutment after implant placement.
  Interventions: Procedure: Placement of dental implant; Procedure: Placement of customized CAD/CAM healing abutment
- Stock Healing Abutments (Active Comparator): Placement of a stock healing abutment after implant placement.
  Interventions: Procedure: Placement of dental implant; Procedure: Placement of stock healing abutment

INTERVENTIONS:
Procedure: Placement of dental implant — Placement of a dental implant on the edentulous ridge
Procedure: Placement of stock healing abutment — Placement of stock healing abutment after implant has been placed on the edentulous ridge
  Arms: Stock Healing Abutments
Procedure: Placement of customized CAD/CAM healing abutment — Placement of customized CAD/CAM healing abutment after implant has been placed on the edentulous ridge
  Arms: Customized Healing Abutments

SUMMARY:
Our long-term goal is to generate evidence for the creation of successful implant restorations and ideal supporting tissues in adequate health by utilizing patient-tailored implant protocols such as the use of customized computer-aided design and computer-aided manufacturing (CAD/CAM) healing abutments. With this study, the investigators intend to recruit patients requiring a single implant placement and implant crown in molar areas. Patients will be randomly assigned to either the control group that will receive standard healing abutments or the test control group that will receive customized CAD/CAM healing abutments. Patients will be followed for six months after the delivery of the implant crowns. The central hypothesis is that the use of customized CAD/CAM healing abutments will demonstrate improved outcomes in terms of hard and soft tissue volume stability and clinical parameters as compared to the use of standard healing abutments.

Aim 1 will measure soft and hard tissue changes around dental implants when customized CAD/CAM healing abutments are utilized as compared to standard healing abutments. Soft tissue stability will be measured utilizing intraoral digital scans, while osseous levels will be measured utilizing CBCT scans. Soft and hard tissue volumetric and linear changes will be measured by digital scan superimposition at the time of crown delivery and 6 months thereafter. Volumetric and linear changes will be compared within each group at different time points and between the test and control group to determine if the use of customized CAD/CAM healing abutments is advantageous in terms of maintaining peri-implant soft and hard tissue stability.

Aim 2 will assess different clinical measurements around dental implants to analyze if the use of customized CAD/CAM healing abutments will demonstrate improved plaque control and peri-implant health as compared to standard healing abutments. Plaque index (PI), gingival index (GI), probing depths (PD), and bleeding on probing (BOP) will be obtained at the time of crown delivery and at 3 and 6 months. Clinical measurements will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will aid in obtaining a natural looking restoration that would result in improved clinical parameters that measure peri-implant health.

Aim 3 will compare the degree of patient satisfaction using a visual analogue scale (VAS) in patients that received an implant restoration following the use of a customized CAD/CAM healing abutment as compared to standard healing abutments. Patients will complete a VAS questionnaire that will evaluate patient perception of pain, esthetics, ability to chew, and ability to clean. Scores will be compared among groups to evaluate if there is a difference in patient-centered outcomes when customized healing abutments are used as compared to standard healing abutments.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Missing a maxillary or mandibular molar that can be replaced with a dental implant
* Sufficient bone volume for standard-sized implants
* Presence of adjacent teeth (mesial and distal)
* No requirement of additional osseous grafting or soft tissue augmentation

Exclusion Criteria:

* Patients <18 years
* Pregnant women
* Active periodontal disease
* Presence of caries or periapical pathology in adjacent teeth
* Use of medications that can impair osseous healing (bisphosphonates, RANKL inhibitors, proton pump inhibitors)
* Current smokers (>10 cigarettes per day)
* Uncontrolled diabetes (HBA1c >8)
* <3mm of keratinized tissue at implant site
* History of head or neck radiation therapy
* History of chemotherapy within the last 4 years
* Uncontrolled alcohol use (more than 4 drinks on any day or more than 14 drinks per week for men and more than 3 drinks on any day or more than 7 drinks per week for women)
* Illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Linear soft tissue changes around dental implants | baseline and 6 months after crown delivery
  Soft tissue linear changes will be measured by digital scan superimposition at the time of crown delivery and 6 months thereafter in millimeters. Linear changes will be compared within each group at different time points and between the test and control group to determine if the use of customized CAD/CAM healing abutments is advantageous in terms of minimizing changes.
Volumetric soft tissue changes around dental implants | baseline and 6 months after crown delivery
  Soft tissue volumetric changes will be measured by digital scan superimposition at the time of crown delivery and 6 months thereafter in cubic millimeters. Volumetric changes will be compared within each group at different time points and between the test and control group to determine if the use of customized CAD/CAM healing abutments is advantageous in terms of minimizing changes.
Linear hard tissue changes around dental implants | baseline and 6 months after crown delivery
  Hard tissue (osseous) linear changes will be measured utilizing a STL file obtained from the CBCT scans. Hard tissue linear changes will be measured by digital superimposition at the time of crown delivery and 6 months thereafter in millimiters. Linear changes will be compared within each group at different time points and between the test and control group to determine if the use of customized CAD/CAM healing abutments is advantageous in terms of minimizing changes.
Volumetric hard tissue changes around dental implants | baseline and 6 months after crown delivery
  Hard tissue (osseous) volumetric changes will be measured utilizing a STL file obtained from the CBCT scans. Hard tissue volumetric changes will be measured by digital superimposition at the time of crown delivery and 6 months thereafter in cubic millimiters. Volumetric changes will be compared within each group at different time points and between the test and control group to determine if the use of customized CAD/CAM healing abutments is advantageous in terms of minimizing changes.
Clinical measurements around implants: Plaque index (PI) | baseline
  Plaque index (PI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall PI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Plaque scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Plaque index (PI) | 3 months after crown delivery
  Plaque index (PI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall PI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Plaque scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Plaque index (PI) | 6 months after crown delivery
  Plaque index (PI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall PI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Plaque scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Gingival Index (GI) | baseline
  Gingival index (GI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall GI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Gingival index scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Gingival Index (GI) | 3 months after crown delivery
  Gingival index (GI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall GI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Gingival index scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Gingival Index (GI) | 6 months after crown delivery
  Gingival index (GI) will be recorded at six sites around the implant crown (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual). Each site will be graded based on a scale from 0 to 3 and the sum of all sites will calculate the overall GI ranging from 0 to 18 (0 being the best outcome possible and 18 the worst outcome possible). Gingival index scores will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Probing depths (PD) | baseline
  Probing depths (PD) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) from the gingival margin to the base of the sulcus around the implant crown. Each site will be measured in millimeters. Probing depths will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Probing depths (PD) | 3 months after crown delivery
  Probing depths (PD) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) from the gingival margin to the base of the sulcus around the implant crown. Each site will be measured in millimeters. Probing depths will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Probing depths (PD) | 6 months after crown delivery
  Probing depths (PD) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) from the gingival margin to the base of the sulcus around the implant crown. Each site will be measured in millimeters. Probing depths will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Bleeding on probing (BOP) | baseline
  Bleeding on probing (BOP) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) around the implant crown. BOP will be recorded as positive if it occurs within 30 seconds of probing and recorded as negative if it does not occur. BOP will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Bleeding on probing (BOP) | 3 months after crown delivery
  Bleeding on probing (BOP) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) around the implant crown. BOP will be recorded as positive if it occurs within 30 seconds of probing and recorded as negative if it does not occur. BOP will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Clinical measurements around implants: Bleeding on probing (BOP) | 6 months after crown delivery
  Bleeding on probing (BOP) will be recorded at six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) around the implant crown. BOP will be recorded as positive if it occurs within 30 seconds of probing and recorded as negative if it does not occur. BOP will be compared between the test and control group to determine if the use of customized CAD/CAM healing abutments will result in improved clinical parameters that measure peri-implant health.
Degree of patient satisfaction | 6 months after crown delivery
  Patients will complete a visual analogue scale (VAS) questionnaire. On a scale from 0 to 10 (0 being the worst outcome possible and 10 the best outcome possible), patients will be asked their perception of pain during the procedure, esthetics, ability to chew and ability to clean. Scores will be compared among groups to evaluate if there is a difference in patient-centered outcomes when customized healing abutments are used as compared to standard healing abutments.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University School of Dental Medicine, Greenville, North Carolina, United States